#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan Amendment 1 for An Open-<br>label, Randomized, Single dose, Crossover, Pivotal<br>Bioequivalence Study of Fixed-dose Combination Tablets of<br>Dolutegravir and Lamivudine versus Dolutegravir and<br>Lamivudine single entities and Food Effect Assessment in<br>Healthy Volunteers |
|---|---|---|
| <b>Compound Number</b> | : | GSK3515864 (GSK1349572+GR109714) |
| <b>Effective Date</b> | : | 28-AUG-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204994
- This RAP is intended to describe the safety, pharmacokinetics (PK), and tolerability analyses required for the study.
- This version of the RAP includes amendment 1 to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | (Clinical Statistics, PAREXEL) | 22-AUG-2017 |
|-----|--------------------------------|-------------|
|-----|--------------------------------|-------------|

#### The Clinical Statistician (or designee) will give final approval:

| (Clinical Statistics, GSK) | 23-AUG-2017 |
|----------------------------|-------------|
|----------------------------|-------------|

#### **Revision Chronology**

| Date | Version |
|---|---|
| 26-JUL-2017 | Original |
| 28-AUG-2017 | Amendment No. 1 |
| Amendment 1 provides clarity that a similar preliminary PK | analysis as was conducted |

Amendment 1 provides clarify that a similar preliminary PK analysis as was conducted following Part 1, will also be performed for Part 2.

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS | PLAN SYNOPSIS | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | Changes<br>Study Ol<br>Study De | s to the Pro<br>bjective(s)<br>esign | TOCOL INFORMATIONtocol Defined Statistical Analysis Pand Endpoint(s) | lan6<br>6 |
| 3. | PLANI<br>3.1.<br>3.2. | Interim A | Analyses | | 9 |
| 4. | ANAL`<br>4.1. | | | 3 | |
| 5. | | | | DATA ANALYSES AND DATA HAI | |
| 6. | STUD<br>6.1. | | | ALYSESd Analyses | |
| 7. | PRIMA<br>7.1. | | cokinetic Ai<br>Overview<br>Drug Con | NALYSESof Planned Pharmacokinetic Analycentration Measuresokinetic Parameters | |
| 8. | SECO<br>8.1. | | nalyses | AL ANALYSESof Planned Analyses | 16 |
| 9. | REFE | RENCES. | | | 18 |
| 10. | APPEI<br>10.1.<br>10.2.<br>10.3.<br>10.4. | Appendi<br>Appendi<br>Appendi<br>Appendi<br>10.4.1.<br>10.4.2. | x 1: Protoc<br>x 2: Data M<br>x 3: Time &<br>x 4: Treatm<br>Treatmen<br>Treatmen<br>10.4.2.1.<br>x 5: Data D<br>Study Tre<br>Baseline I | ol Deviation Management | |

#### CONFIDENTIAL

| | | 10.5.2.2. | Derivations and Handling of Missing Baseline | |
|---|---|---|---|---|
| | | | Data | 26 |
| | 10.5.3. | Reporting I | Process & Standards | 26 |
| 10.6. | Appendix | 6: Derived | and Transformed Data | 29 |
| | 10.6.1. | General | | 29 |
| | 10.6.2. | Study Popu | ulation | 29 |
| | 10.6.3. | | | |
| 10.7. | Appendix | 7: Prematu | ure Withdrawals & Handling of Missing Data | 31 |
| | 10.7.1. | Premature | Withdrawals | 31 |
| | 10.7.2. | Handling of | f Missing Data | 31 |
| | | 10.7.2.1. | Handling of Missing Dates | 31 |
| | | 10.7.2.2. | Handling of PK Concentration Data | 32 |
| 10.8. | Appendix | 8: Values | of Potential Clinical Importance | 33 |
| | 10.8.1. | | Values | |
| | 10.8.2. | ECG | | 33 |
| | 10.8.3. | Vital Signs | | 33 |
| 10.9. | Appendix | 9: Model C | Checking and Diagnostics for Statistical | |
| | 10.9.1. | Statistical A | Analysis Assumptions | 34 |
| 10.10. | | | viations & Trade Marks | |
| | 10.10.1. | Abbreviation | ons | 35 |
| | 10.10.2. | Trademark | S | 36 |
| 10.11. | Appendix | 11: List of | Data Displays | 37 |
| | 10.11.1. | Data Displa | ay Numbering | 37 |
| | 10.11.2. | Mock Exan | nple Referencing | 37 |
| | 10.11.3. | Study Popu | ulation Tables | 38 |
| | 10.11.4. | Pharmacok | kinetic Tables | 39 |
| | 10.11.5. | Pharmacok | kinetic Figures | 51 |
| | 10.11.6. | Safety Tab | les | 60 |
| | 10.11.7. | ICH Listing | S | 62 |
| | 10.11.8. | Non-ICH Li | istings | 65 |
| 10.12. | | | ole Mock Shells for Data Displays | |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the Clinical Pharmacology |
| Protocol | Study Report for Protocol 204994 This RAP is based on the original protocol (Dated: 12-JAN-2017) of study |
| Protocol | GSK204994 (GSK Document No.: 2016N286215_00) and protocol amendment 1 (Dated: 07-FEB-2017) of study GSK204994 (GSK Document No.: 2016N286215_01) |
| Primary<br>Objective | To evaluate the bioequivalence (BE) of fixed-dose combination (FDC) tablet formulation(s) of DTG 50 mg and 3TC 300 mg versus coadministration of the separate tablet formulations of DTG 50 mg plus 3TC 300 mg, in the fasted state. |
| Primary<br>Endpoint | Plasma DTG and 3TC $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , and $C_{max}$ . |
| Study<br>Design | This is a single-center, open-label, randomized, two-part study (if Part 2 is conducted) |
| | Part 1, Bioequivalence and Food Effect (FD) with Monolayer FDC Tablet Part 1 of the study will be a randomized, open-label, 2-period, single-dose, crossover study in 76 healthy adult subjects to achieve at least 70 evaluable subjects. The first 16 subjects who complete the first two treatment periods, and consent to continue, will return for a third treatment period and receive a single dose of the FDC tablet formulation administered with a high fat meal. Treatment Period 1 A: Reference treatment DTG + 3TC Or B: FDC formulation Part 2 Bioequivalence and Food Effect with Bilayer FDC Tablet |
| | Part 2, Bioequivalence and Food Effect with Bilayer FDC Tablet Part 2 of the study, incorporating the bilayer FDC formulation, will only be conducted if a suitable formulation is available. Part 2 of the study will be conducted, similarly to Part 1. |
| | Treatment Period 1 A: Reference treatment DTG + 3TC Or C: FDC formulation Solve A Treatment Period 2 A: Reference treatment DTG + 3TC Or C: FDC formulation Solve A Treatment Period 2 A: Reference treatment DTG + 3TC Or C: FDC formulation With high fat meal |
| Planned<br>Analyses | Interim analyses are detailed within Section 3.1. The Good along a development of the control of the cont |
| | The final planned analyses will be performed after the completion of the study and final datasets authorization, i.e. when database freeze |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| | (DBF) is declared. |
| Analysis | Screening Population |
| Population | Safety Population |
| | PK Plasma Concentration Population |
| | PK Parameter BE Summary Population |
| | PK Parameter FD Summary Population |
| Hypothesis | <ul> <li>The first two treatment periods of each part of this study are designed to test the BE of FDC tablets of DTG and 3TC (test treatment) relative to coadministered DTG plus 3TC (reference treatment) all under fasting condition:</li> <li>H(0): μ(test)/μ(reference) &lt; 0.800 or μ(test)/μ(reference) &gt; 1.250, i.e., treatments are not bioequivalent.</li> <li>Versus</li> <li>H(1): 0.800 ≤ μ(test)/μ(reference) ≤ 1.250 i.e., treatments are bioequivalent.</li> </ul> |
| | Food Effect: No formal hypothesis will be tested and an estimation approach will be used to evaluate the effect of food on the FDC tablet(s). |
| Primary<br>Analyses | Following loge-transformation, AUC <sub>(0-∞)</sub> , AUC <sub>(0-t)</sub> , C <sub>max</sub> from the first two treatment periods for BE will be separately analyzed for each analyte using a mixed effects model. Point estimates and their associated 90% confidence intervals (CIs) will be provided for the ratios of PK parameters between test and reference treatments on the original scale. |
| Secondary<br>Analyses | PK data will be presented in graphical and/or tabular form and will be summarized descriptively. |
| | <ul> <li>Following loge-transformation, AUC<sub>(0-24)</sub>, C<sub>24</sub>, CL/F and t<sub>1/2</sub> from the first two treatment periods for BE, and AUC<sub>(0-∞)</sub>, AUC<sub>(0-t)</sub>, C<sub>max</sub>, CL/F, AUC<sub>(0-24)</sub>, C<sub>24</sub>, t<sub>1/2</sub> from the third treatment period (food effect) will be analysed similarly using a mixed effects model.</li> <li>T<sub>max</sub> and t<sub>lag</sub> of DTG and 3TC will be separately analyzed with the nonparametric Wilcoxon matched pair method to compute point estimates and associated 90% CIs for the median differences.</li> <li>Safety data will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. No formal statistical analysis of the safety data will</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Except for the addition of a similar preliminary PK analysis for Part 2 as was conducted for Part 1, there were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 1 [Dated: 07-FEB-2017].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the bioequivalence of FDC tablet formulation(s) of DTG 50 mg and 3TC 300 mg versus co-administration of the separate tablet formulations of DTG 50 mg plus 3TC 300 mg, in the fasted state. | Plasma DTG and 3TC $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , and $C_{max}$ . |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To characterize the PK profile of single dose of FDC tablet formulation(s) of DTG 50 mg and 3TC 300 mg versus coadministration of the separate tablet formulations of DTG 50 mg plus 3TC 300 mg, in the fasted state</li> <li>To evaluate the food effect on FDC tablet formulation(s) of DTG 50 mg and 3TC 300 mg</li> </ul> | <ul> <li>Plasma DTG and 3TC t<sub>lag</sub>, t<sub>max</sub>, t, t<sub>½</sub>, λz, %AUC<sub>ex</sub>, AUC<sub>(0-24)</sub>, CL/F and Vz/F, C<sub>t</sub>, and C<sub>24</sub></li> <li>Plasma DTG and 3TC AUC<sub>(0-∞)</sub>, AUC<sub>(0-t)</sub>, C<sub>max</sub>, t<sub>lag</sub>, t<sub>max</sub>, t, t½, λz, %AUC<sub>ex</sub>, AUC<sub>(0-24)</sub>, CL/F and Vz/F, C<sub>t</sub>, and C<sub>24</sub>.</li> </ul> |
| To assess the safety and tolerability from single dose administration of the combination of DTG 50 mg, 3TC 300 mg in healthy volunteers either fasted or with a high fat meal. ALC as a great under the plasma concentration time curve from the curve from the curv | Safety and tolerability parameters as assessed by change from baseline in vital signs (BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests |

AUC<sub>(0-t)</sub>= area under the plasma concentration time curve from time zero to the last quantifiable time point

AUC<sub>(0-∞)</sub>= area under the plasma concentration time curve from time zero to infinity

AUC<sub>(0-24)</sub>= area under the plasma concentration time curve from time zero to 24 hours

%AUC<sub>ex</sub>=% of AUC<sub>(0-∞)</sub> that was extrapolated

C<sub>max</sub>= maximum observed concentration

 $t_{\text{max}}$ = time of maximum observed concentration

C<sub>24</sub>= concentration at 24h post-dose

C<sub>t</sub> = last quantifiable concentration

PK = Pharmacokinetic

t = time of last quantifiable concentration

t<sub>lag</sub>= absorption lag time

λz=apparent elimination rate constant

 $t_{1/2}$  = the elimination half-life

CL/F = apparent oral clearance

Vz/F= apparent oral volume of distribution

# 2.3. Study Design



| Overview of S | Study Design and Key Featur | es | | |
|---|---|---|---|---|
| Treatment | Subjects will be randomized | to one of the fol | lowing two seq | uences in Part 1 |
| Assignment | | | | |
| | Sequences | Period 1 | Period 2 | Period 3 |
| | | Bioequivalen<br>Crossove | | Food effect <sup>a</sup> |
| | Part 1 | | | 101 |
| | A/B, n=38 | Α | В | B Fed |
| | B/A, n=38 | В | Α | (n=16) |
| | Part 2 (if conducted) | | • | |
| | A/C, n=38 | Α | С | C Fed |
| | C/A, n=38 | С | Α | (n=16) |
| | Treatment A = DTG 50 mg tablet | (clinical image) plu | s a single EPIVIR | 300 mg tablet |
| Interim | Treatment B = DTG 50 mg/3TC 300 mg FDC monolayer formulation (Product code AH) Treatment C = DTG 50 mg/3TC 300 mg FDC bilayer formulation (Product code TBD) a. first 16 subjects who complete the two treatment periods, and consent to continue to complete period 3 in each part Subjects will be administered the 1 <sup>st</sup> treatment in the sequence in the 1 <sup>st</sup> period; the 2 <sup>nd</sup> treatment in the sequence in the 2 <sup>nd</sup> period; • Each treatment will be administered in the fasted state after at least 10 hours of fasting in the first two treatment periods. • Each treatment will be administered with a high fat meal in the third treatment period. Following completion of Part 1, preliminary PK data from Part 1 will be | | | |
| Analysis | analyzed. The point estimate for the ratio of the geometric geometric mean of the refere AUC <sub>(0-t)</sub> , and C <sub>max</sub> for both D A similar preliminary PK and also be performed for Part 2. Phase III study. An independ perform the preliminary PK and perform the performance performa | s and correspond<br>mean of the test<br>nce treatments, p<br>OTG and 3TC.<br>alysis as was con<br>The result will b<br>lent statistics and | ling 90% CIs we treatment (more u(test)/µ(referent ducted following used for plant programming | rill be constructed nolayer) to the nce) for $AUC_{(0-\infty)}$ , ng Part 1, will ning a future |

# 2.4. Statistical Hypotheses

The first two treatment periods of each part of this study are designed to test the bioequivalence of FDC tablets of DTG and 3TC (test treatment) relative to coadministered DTG plus 3TC (reference treatment) all under fasting condition. The null hypothesis is that the true ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment,  $\mu(\text{test})/\mu(\text{reference})$ , for each primary PK endpoint, is either less than 0.800 or greater than 1.250. The alternate hypothesis is that the true ratio of the test treatment geometric mean to the reference treatment geometric mean is greater than or equal to 0.800 and less than or equal to 1.250. Symbolically, this

is expressed as follows:

- H(0):  $\mu(\text{test})/\mu(\text{reference}) < 0.800$  or  $\mu(\text{test})/\mu(\text{reference}) > 1.250$ , i.e., treatments are not bioequivalent versus
- H(1):  $0.800 \le \mu(test)/\mu(reference) \le 1.250$  i.e., treatments are bioequivalent. For each PK parameter designated as a primary endpoint (see Section 2.2), a two one-sided t-test (TOST) procedure (Schiurmann, 1987) with  $\alpha$ =0.05 for each one-sided test will be used to test this set of hypotheses. This is equivalent to requiring that a 90% interval for the true ratio of test to reference geometric means falls entirely within the range of 0.800 to 1.250. To declare bioequivalence of FDC tablet DTG and 3TC to coadministered DTG plus 3TC, the primary PK endpoints for both analytes should demonstrate bioequivalence.

For the food effect portion(s), no formal hypothesis will be tested and an estimation approach will be used to evaluate the effect of food on the FDC tablet.

#### 3. PLANNED ANALYSIS

## 3.1. Interim Analyses

Following completion of Part 1, preliminary PK data from Part 1 will be analyzed. The point estimates and corresponding 90% CIs will be constructed for the ratio of the geometric mean of the test treatment (monolayer) to the geometric mean of the reference treatments,  $\mu(\text{test})/\mu(\text{reference})$  for  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ , and  $C_{\text{max}}$  for both DTG and 3TC.

A similar preliminary PK analysis as was conducted following Part 1, will also be performed for Part 2. This is simply bringing forward a part of the planned end of study analysis to pre-DBF, but after all subjects have completed the trial, in order to expedite decision making. The PK parameter data for the preliminary analysis will be based on the nominal sampling times.

The result will be used for planning a future Phase III study. An independent statistics and programming team will perform the preliminary PK analyses for both part1. As the PK data are analyzed separately for each part of the study, there will be no adjustments for multiplicity.

# 3.2. Final Analyses

| Analysis | Details |
|---|---|
| Final Analyses | Final analyses will be performed after the completion of the study and final database authorization. |

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screening<br>Population | All subjects who signed the consent form will be included in this population. | Subject Disposition |
| Safety<br>Population | All subjects who enrolled in the study and received at least one dose of study drug will be included in the Safety Population. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic (PK) Plasma Concentration | The PK Plasma Concentration<br>Population will include all<br>subjects who undergo plasma PK<br>sampling and have evaluable PK<br>assay results for DTG or 3TC. | <ul> <li>PK concentration listings,</li> <li>calculating PK parameters,</li> <li>PK parameter listings</li> <li>plotting of the individual concentration-time profiles</li> </ul> |
| Pharmacokinetic<br>(PK) Parameter<br>BE Summary | The PK Parameter BE Summary Population will include all subjects who have evaluable PK parameters for both analytes and for both Period 1 and Period 2. Data from subjects who vomit within 4 hours of study drug administration will not be considered as evaluable. | <ul> <li>PK concentration summary</li> <li>PK parameter summary and figure</li> <li>Statistical analysis of parameter data</li> <li>Excluded subjects will be included in footnotes for summary tables</li> </ul> |
| Pharmacokinetic<br>(PK) Parameter<br>FD Summary | The PK Parameter FD Summary Population will include subjects who participate in the food effect part of study, and have evaluable PK parameters for both fed and fasted administration of the FDC tablet formulation. Data from subjects who vomit within 4 hours of study drug administration will not be considered as evaluable. | <ul> <li>PK concentration summary</li> <li>PK parameter summary and figure</li> <li>Statistical analysis of parameter data</li> <li>Excluded subjects will be included in footnotes for summary tables</li> </ul> |

#### NOTES:

- Please refer to Appendix 11 which details the population to be used for each display being generated.
- Additional PK concentration and parameter summary tables will be provided by using the PK plasma concentration
  population if there are subjects with only 1 period PK data or subjects who vomit.

#### 4.1. Protocol Deviations

- All protocol deviations will be listed with flags to indicate whether a PD is important and results in exclusion from the analysis population.
- Important deviations will also be summarized, reported in the study report (Please refer to Appendix 1: Protocol Deviation Management).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised in the protocol deviations dataset.
  - o This dataset will be the basis for the listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Data Management |
| 10.3 | Appendix 3: Time & Events |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses. |
| 10.10 | Appendix 10: Abbreviations and Trade Marks |
| 10.11 | Appendix 11: List of Data Displays |
| 10.12 | Appendix 12: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data I | Displays Ger | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomization | • | | |
| Randomization | | | Y |
| <b>Subject Disposition</b> | | | |
| Subject Disposition | | Y | |
| Reasons for Screening Failures | | | Y <sup>[1]</sup> |
| Reasons for Withdrawals | | | Y |
| Important <sup>[3]</sup> Protocol Deviations | | Y | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Subjects Excluded from Analysis Populations | | | $Y^{[2]}$ |
| Demography | | | |
| Demographics Characteristics | | Y | Y |
| Race & Racial Combinations | | Y | Y |
| Concomitant Medications | | | |
| Concomitant Medication | | | Y |

#### NOTES:

- Y = Yes display generated.
- 1. Conditional displays, if data is available listing will be generated.
- 2. Listing of subjects excluded from any population will be generated only.
- 3. All protocol deviations will be listed, with important protocol deviations summarized.

#### 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Pharmacokinetic Analyses

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of, Clinical Pharmacology Sciences and Study Operations (CPSSO) data management, GlaxoSmithKline.

The merge of PK concentration data, randomization and CRF data will be performed by Study Data Tabulation Model (SDTM) programmer at Quintiles and the analysis PK

concentration dataset and WinNonLin files will be created by statistics and programming, PAREXEL, under the direct auspices of statistics and programming, Quantitative Sciences (QSci), GlaxoSmithKline.

Derivation of pharmacokinetic parameters will be performed by Clinical Pharmacology Modelling & Simulation (CPMS), QSci, GlaxoSmithKline.

Statistical Analysis of pharmacokinetic parameters will be performed by statistics and programming, PAREXEL, under the direct auspices of statistics and programming, QSci, GlaxoSmithKline.

#### 7.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "PK Plasma Concentration" or "PK Parameter BE or FD Summary' populations, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

| Endpoints | 1 | Untransformed | | | L | og <sub>e</sub> -Tra | nsforme | d |
|---|---|---|---|---|---|---|---|---|
| | Sumn | Summary | | ridual | Sum | mary | Indiv | ridual |
| | F | T | F | L | F | T | F | L |
| Plasma Drug<br>Concentrations | Y [1] [2] | Y | Y [1] | Y | | | | |
| Derived PK Parameters | | Y | $Y^{[3]}$ | Y | $Y^{[4]}$ | Y | Y | |
| Statistical Analysis PK<br>Parameters | | | | | Y <sup>[5]</sup> | Y | | Y <sup>[6]</sup> |

Table 3 Overview of Planned Pharmacokinetic Analyses

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- T<sub>max</sub> and t<sub>lag</sub> are not log transformed.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Mean (+SD) and Median plots will be generated.
- 3. Comparative Plot of Individual DTG and 3TC Plasma PK Parameter versus treatments
- 4. Treatment Comparative Plot of adjusted geometric mean (95% CI) with Individual Subject Plasma PK Parameters will be generated.
- Geometric Mean Treatment Ratio and 90% CI of DTG and 3TC Plasma PK Parameters will be generated.
- Supportive SAS Output from Statistical Analysis of Loge-transformed DTG and 3TC Plasma PK Parameters

#### 7.1.2. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

#### 7.1.3.1. Deriving Pharmacokinetic Parameters

- PK analyses will be the responsibility of the CPMS department within GSK or their designee. Plasma DTG and 3TC concentration-time data will be analyzed by non-compartmental methods according to current working practices and using Phoenix WinNonlin 6.3 or higher. Calculations will be based on the actual sampling times recorded during the study and based on nominal sampling times. From the plasma concentration-time data, the following PK parameters will be determined, as data permit: C<sub>max</sub>, T<sub>max</sub>, AUC<sub>(0-t)</sub>, AUC<sub>(0-∞)</sub>, AUC<sub>(0-24)</sub>, t<sub>1/2</sub>, t<sub>lag</sub>, C<sub>24</sub>, C<sub>t</sub>, λz, %AUC<sub>ex</sub>, Vz/F, t and CL/F.
- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- Non-compartmental analysis will be performed in accordance with GSK PK Guidance document GUI 51487.
- Two sets of PK parameters will be derived for each subject, analyte and treatment: one set based on actual sampling times and one set based on nominal times.
- Pharmacokinetic parameters described in Table 4 will be determined from plasma concentration-time data, as data permit.

Refer Appendix 7 Section 10.7.2.2 for handling of PK Concentration data.

Table 4 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| $\mathrm{AUC}_{(0-\infty)}$ | Area under the concentration-time curve from time zero extrapolated to infinity |
| AUC <sub>(0-t)</sub> | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C <sub>t</sub> ) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC <sub>t</sub> (%) | Percent of the area measured by $AUC_{(0-t)}$ relative to the extrapolated $AUC_{(0-\infty)}$ |
| AUC <sub>(0-24)</sub> | Area under the plasma concentration time curve from time zero to 24 hours |
| %AUC <sub>ex</sub> | % of $AUC_{(0-\infty)}$ that was extrapolated |
| C <sub>24</sub> | Drug concentration at 24 hours post-dose |
| C <sub>max</sub> | Maximum observed concentration, determined directly from the concentration-time data. |
| $C_{t}$ | last quantifiable concentration |
| t | time of last quantifiable concentration |
| $T_{\text{max}}$ | Time to reach C <sub>max</sub> , determined directly from the concentration-time data. |
| tlag | Lag time before observation of drug concentrations in sampled matrix |

| Parameter | Parameter Description |
|---|---|
| λz | Apparent elimination rate constant |
| t1/2 | Apparent terminal half-life will be calculated as: $t_{1/2} = \ln 2 / \text{Lambda}_z$ (NOTE: Lambda_z is the terminal phase rate constant). |
| CL/F | The apparent oral clearance (CL/F) will be calculated as CL/F = $Dose/AUC_{(0-\infty)}$ |
| Vz/F | Apparent oral volume of distribution |

#### 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

Two sets of bioequivalence assessments and food effect will be performed based on:

- PK parameters derived based on actual sampling times
- PK parameters derived based on nominal sampling times For each of the parameters  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ ,  $AUC_{(0-24)}$ ,  $C_{max}$ ,  $C_{24}$ ,  $C_t$ , CL/F and  $t_{1/2}$ , the following summary statistics will be calculated and tabulated by treatment (dose):
- Untransformed Data: N, n, arithmetic mean, %CV, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, and maximum.
- **Log**<sub>e</sub>-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of log<sub>e</sub>-transformed data and %CVb

For %AUC<sub>ex</sub>,  $T_{max}$ ,  $t_{lag}$ ,  $\lambda z$ , t, and Vz/F, the summary statistics specified for untransformed data above will be generated.

PK data will be listed and may be presented in graphical form and will be summarized descriptively. All PK data will be stored in the Archives, GlaxoSmithKline R& D.

Statistical analyses of the PK parameter data will be the responsibility of Clinical Statistics, GlaxoSmithKline or their designee.

The PK parameters for DTG and 3TC (except  $T_{max}$  and  $t_{lag}$ ) will be  $log_e$ -transformed and separately analyzed using a mixed effects model. For the analysis of bioequivalence, the model will include fixed effect terms for period and treatment. Subject will be treated as a random effect in the model. For the analysis of food effect, the model will include a fixed effect term for treatment (fed versus fasted) and a random effect term for subject. Point estimates and their associated 90% CIs will be constructed for the differences in PK parameter values between test and reference treatments for the treatment comparisons. The point estimates and their associated 90% CIs will then be back-transformed to provide point estimates and 90% CIs for the ratios of PK parameters between test and reference treatments.

T<sub>max</sub> and t<sub>lag</sub> of DTG and 3TC will be separately analyzed with the non-parametric Wilcoxon matched pair method to compute point estimates and associated 90% confidence intervals for the median differences between test and reference treatments.

#### **Primary and Secondary Comparisons of Interest**

| | DTG or 3TC<br>PK Parameter | Test | Reference | Assessment |
|---|---|---|---|---|
| | | Treatment B | Treatment A | |
| Primary | $AUC_{(0-\infty)},\ AUC_{(0-t)},\ C_{max},$ | Treatment C (if Part 2 is conducted) | Treatment A | Bioequivalence |
| | | Treatment B | Treatment A | |
| | CL/F, AUC <sub>(0-24)</sub> , C <sub>24</sub> , t <sub>1/2</sub> | Treatment C (if Part 2 is conducted) | Treatment A | Bioequivalence |
| Secondary | $AUC_{(0-\infty)},AUC_{(0-t)},C_{max},$ | Treatment B Fed | Treatment B<br>Fasted | |
| | CL/F, AUC <sub>(0-24)</sub> , C <sub>24</sub> , t <sub>1/2</sub> | Treatment C Fed (if Part 2 is conducted) | Treatment C<br>Fasted | Food Effect |

Estimates of within-subject variability for  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ ,  $C_{max}$ , CL/F,  $AUC_{(0-24)}$ ,  $C_{24}$ ,  $t_{1/2}$  will also be provided, where  $CVw(\%) = SQRT(exp(MSE) - 1) \times 100$  and MSE is the residual mean squared error from the model.  $CV_w$  represents a pooled measure of within-subject variability across the treatments A and B or A and C (if Part 2 is conducted).

Comparative Plot of Individual subject DTG and 3TC Plasma PK Parameter Versus Treatment will be generated.

Treatment Comparative Plots of adjusted geometric mean (95% CI) with Individual Subject Plasma PK Parameters  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ ,  $C_{max}$ , CL/F,  $AUC_{(0-24)}$ ,  $C_{24}$ ,  $t_{1/2}$  will be generated.

Plots will also be provided showing the adjusted geometric mean ratio of test to reference treatment for  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ ,  $C_{max}$ , CL/F,  $AUC_{(0-24)}$ ,  $C_{24}$ ,  $t_{1/2}$  with 90% CIs.

The SAS output from the statistical models and the assessment of assumptions underlying the models will be included in a listing of supportive SAS output.

Additional PK displays for Canada specific submission requirements will also be provided.

#### 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Safety Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

#### 8.1.1. Overview of Planned Analyses

Table 5 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Endpoint | | Abs | olute | | Cha | Change from Baseline | | |
|---|---|---|---|---|---|---|---|---|
| _ | Sum | mary | Indiv | /idual | Sumi | mary | Indi | vidual |
| | T | F | F | L | T | F | F | L |
| Exposure | | | | | | | | |
| Exposure | | | | Y | | | | |
| Adverse Events | | | | | | | | |
| All AE's | Y | | | Y | | | | |
| Serious AE's | Y | | | Y | | | | |
| Drug Related AEs | Y | | | Y | | | | |
| Withdrawal AE's | Y | | | Y | | | | |
| Relationship Between | | | | Y | | | | |
| System Organ Class And | | | | | | | | |
| Verbatim Text | | | | | | | | |
| Subject Numbers for | | | | Y | | | | |
| Individual AEs | | | | | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Y | | | | Y | | | |
| Hematology | Y | | | | Y | | | |
| Abnormal Clinical | | | | Y | | | | |
| Chemistry | | | | | | | | |
| Abnormal Hematology | | | | Y | | | | |
| Abnormal Urinalysis | | | | Y | | | | |
| ECG's | | | | | | | | |
| ECG Findings | Y | | | | | | | |
| ECG Values | Y | | | | | | | |
| ECG Values Outside the | | | | Y | | | | |
| PCI Range | | | | | | | | |
| All ECG Values for | | | | Y | | | | |
| Subjects with a Value of | | | | | | | | |
| PCI | | | | | | | | |
| Abnormal ECG Findings | | | | Y | | | | |
| Vital Signs | | | | | | | | |
| Vitals Values | Y | | | | Y | | | |
| Vital Signs Measurements | | 1 | | Y | Y | | | |
| Outside the PCI Range | | | | | | | | |
| All Vital Signs for Subjects | | | | Y | | | | |
| with Values of PCI | | | | | | | | |

## NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 9. REFERENCES

GlaxoSmithKline Document Number 2016N286215\_00: An Open-label, Randomized, Single dose, Crossover, Pivotal Bioequivalence Study of Fixed-dose Combination Tablets of Dolutegravir and Lamivudine versus Dolutegravir and Lamivudine single entities and Food Effect Assessment in Healthy Volunteers. Effective Date: 12-JAN-2017

GlaxoSmithKline Document Number 2016N286215\_01: An Open-label, Randomized, Single dose, Crossover, Pivotal Bioequivalence Study of Fixed-dose Combination Tablet(s) of Dolutegravir and Lamivudine versus Dolutegravir and Lamivudine single entities and Food Effect Assessment in Healthy Volunteers Effective Date: 07-FEB-2107

Schiurmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. *J Pharmacokinetics Biopharm* 1987; 15:657-679.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5 Conventions | : General Considerations for Data Analyses & Data Handling |
| Section 10.2 | Appendix 2: Data Management |
| Section 10.3 | Appendix 3: Time and Events |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | <ul> <li>Appendix 5: Data Display Standards &amp; Handling Conventions</li> <li>Study Treatment &amp; Sub-group Display Descriptors</li> <li>Baseline Definitions &amp; Derivations</li> <li>Reporting Process &amp; Standards</li> </ul> |
| Section 10.6 | <ul> <li>Appendix 6: Derived and Transformed Data</li> <li>General</li> <li>Study Population</li> <li>Safety</li> <li>Pharmacokinetic</li> </ul> |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data General Study Population & Safety |
| Section 10.8 | <ul> <li>Appendix 8: Values of Potential Clinical Importance</li> <li>Laboratory Values</li> <li>ECG</li> <li>Vital Signs</li> </ul> |
| Section 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP A | ppendices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |
| Section 10.12 | Appendix 12: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management

A subject meeting any of the following criteria will be excluded from the PK Parameter BE and/or FD Summary Population:

| Number | Exclusion Description |
|---|---|
| 01 | Failure of any inclusion/exclusion criteria, but subject is still enrolled |
| 02 | A subject with emesis occurring within 4 hours of the dose |

# 10.2. Appendix 2: Data Management

| Data Type | Source | Format | Planned Date of | Responsibility |
|---|---|---|---|---|
| | | of Data | Final File <sup>1</sup> | |
| Safety | Database | SDTM | DBF | CPSSO |
| PK<br>Concentration | SMS2000 data files | dat file | DBF | BIB/BESM |
| PK<br>Concentration<br>(ADPC),<br>WNL File | PK concentration<br>data (SDTM PC),<br>exposure (EX) and<br>demography (DM)<br>datasets <sup>2</sup> | ADaM,<br>CSV file | DBF + 5 Days <sup>1</sup> | QSci |
| PK<br>Parameters | WNL file | CSV file | PK Concentration,<br>WNL file + 5<br>Days | CPMS |

<sup>1.</sup> Provided SDTM PC, EX and DM are in time and clean

PK concentration data is released via SMS2000 by Bioanalysis, Immunogenicity and Biomarkers (BIB)/Bioanalytical External Study Monitors (BESM) and the SDTM PC contains date/times and PK sample ID

# 10.3. Appendix 3: Time & Events

# **Screening Assessments**

| Visit Window (relative to Day 1) | Day -30 to -2 | Notes |
|---|---|---|
| Informed Consent | Х | |
| Demographics | X | |
| Physical examination height, weight and BMI | X | |
| Medical/medication/ history | X | Medical/medication/drug and alcohol history will be recorded at screening, and updated at admission. |
| Urine drug / Cotinine and Breathalyzer screening | X | |
| 12-lead ECG and Vital Signs | X | |
| Serum or urine hCG test (female subjects only) | X | <ul> <li>See inclusion Protocol criterion #6.</li> <li>Performed at site standard procedure.</li> </ul> |
| FSH and estradiol (women) | X | |
| HIV, Hep B and Hep C Screen | X | |
| Hematology/Chemistry/Urinalysis tests | X | |

## **Treatment Period Assessments**

| | All Dosing Periods | | | | | | | ď | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Day -1 | Day 1 | | | Day<br>2 | Day<br>3 | Day<br>4 | Follow-up | Notes | |
| | | Pre-<br>dose | 0 hr | | Post Dose | - | 48 hr | 72 hr | E | Day -1 of Periods 2 to 3 may be the same day as Day 6 of prior periods |
| Admission to Unit | Χ | | | | | | | | | |
| Discharge | | | | | | | Х | | | |
| Outpatient Visit | | | | | | | | Χ | Χ | Follow-up visit will occur 7 to 14 days post last dose. |
| 12-lead ECG | Х | | | | | | | | | Single ECGs will be collected at Screening and on Day-1 of Period 1 only. Additional ECGs may be performed at the discretion of the investigator. |
| Vital signs | Х | Χ | | At 4 | 4 hours post-dose | Χ | Χ | Χ | Χ | Single measurements performed at all time points. |
| Brief Physical Exam | Χ | | | | | | | | | Brief examinations may be made full examinations and |
| Urine Drug/ Cotinine and Breathalyzer | Х | | | | | | | | | <ul> <li>laboratory procedures may be repeated, if needed, at the discretion of the Investigator.</li> <li>Illicit Drug/Alcohol/Cotinine/pregnancy screening will be performed in accordance with the sites' standard practice.</li> <li>Clinical laboratory tests – see Protocol Table 5.</li> </ul> |
| Pregnancy test | Χ | | | | | | | | Х | |
| Clinical laboratory tests | Χ | | | | | | | | Х | |
| Dosing | | | Х | | | | | | | Subject will be dosed while in the seated position. |
| Pharmacokinetic Sampling | | Х | | | ect at 0.25, 0.5, 0.75, 1<br>5, 6, 8, 12, 16, 24, an<br>dose | | | Х | | Pre-dose (within 15 minutes prior to dosing). 4 hour post dose sample must be taken <u>prior to</u> provision of food. Permitted window for the collection of PK sample at each time point will be specified in BioPacket. |
| Meals – (Treatment periods 1 and 2) | | sted from 10 hours prior to<br>osing to 4 hours post-dose | | Standard for the study center | | | | See also Protocol Section 6.10.1.1 | | |
| Meals - Treatment Period 3<br>(Fed Conditions only) | Fasted from 10 hours prior to<br>test meal and dosing then<br>through 4 hours post-dose | | Standard for the | study ce | nter | | | Entire meal to be consumed in 25 minutes or less and dosing will be administered 30 minutes after the start of the meal. See also Protocol Section 6.10.1.2 | | |
| Adverse Events | Χ | X <b>←</b> ===========X=====X | | | <b>&gt;</b> | Χ | | | | |
| Concomitant medications | Х | <b>←==</b> | ===== | ====== | ======X====== | ===== | ====== | == <b>→</b> | Χ | |

# 10.4. Appendix 4: Treatment States and Phases

#### 10.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the start and/or stop date/time of the study treatment.

| Treatment<br>Phase | Definition |
|---|---|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time < Date/Time ≤ [Study Treatment Stop Date/Time + 3 Days] |
| Post-Treatment | Date/Time > [Study Treatment Stop Date/Time + 3 Days] |

#### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date/time of the study treatment.

#### 10.4.2.1. Treatment States for AE Data

| Treatment<br>State | Definition |
|---|---|
| Pre-Treatment | AE Start Date/Time < Study Treatment Start Date/Time |
| On-Treatment | If AE onset date/time is on or after treatment start date/time & 3 or fewer days after the treatment stop date/time Study Treatment Start Date/Time ≤ AE Start Date/Time ≤ [Study Treatment Stop Date/Time + 3] |
| Post-<br>Treatment | If AE onset date/time is more than 3 days after the treatment stop date/time AE Start Date/Time > [Study Treatment Stop Date/Time + 3] |
| Onset Time<br>Since First<br>Dose<br>(Days) | If Treatment Start Date/Time > AE Onset Date/Time = AE Onset Date - Treatment Start Date If Treatment Start Date/Time ≤ AE Onset Date/Time = AE Onset Date - Treatment Start Date +1 Missing otherwise |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF |

#### **NOTES:**

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | |
|---|---|---|
| RandAll NG Data Displays for Reporting | | |
| Code | Description | Description |
| A | DTG 50mg plus EPIVIR 300mg | A |
| В | DTG 50mg and 3TC 300mg FDC monolayer | В |
| С | DTG 50mg and 3TC 300mg FDC bilayer | С |
| B_Fed <sup>[1]</sup> | DTG 50mg and 3TC 300mg FDC monolayer fed | B_Fed |
| C_Fed <sup>[1]</sup> | DTG 50mg and 3TC 300mg FDC bilayer fed | C_Fed |

<sup>[1]</sup> Treatments B Fed and C Fed are assigned.

**NOTES:** Add the following footnote for treatment description.

A: DTG 50mg plus EPIVIR 300mg

B: DTG 50mg and 3TC 300mg FDC monolayer

C: DTG 50mg and 3TC 300mg FDC bilayer

B\_Fed: DTG 50mg and 3TC 300mg FDC monolayer fed

C\_Fed: DTG 50mg and 3TC 300mg FDC bilayer fed

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

For all endpoints (except as noted in the table) the baseline value will be the latest predose assessment.

Table 6 Baseline Definitions

| Dougneton | Study Asses | ssments Co<br>Baseline | Baseline Used in | |
|---|---|---|---|---|
| Parameter | Screening | Day -1 | Day 1<br>(Pre-Dose) | Data Display |
| Safety | | | | |
| Lab | X | X | | Day -1 |
| Vital Signs (blood pressure, and pulse rate) | X | X | X | Day 1 (Pre-Dose) for each Period |

#### 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### **NOTES:**

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.5.3. Reporting Process & Standards

| Software | |
|---|---|
| • The currently supported versions of SAS and S-Plus software will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259-HARP PROD-US |
| HARP Area | : \ARPROD\GSK1349572\mid204994\Final |
| QC Spreadsheet : \ARWORK\GSK1349572\mid204994\Final\Documents | |
| Analysis Datasat | Analysis Datasets |

#### **Analysis Datasets**

Reporting Process

 Analysis datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) standards (SDTM IG Version 3.1.3 & Analysis Data Model (ADaM) Implementation Guide (ADaM IG) Version 1.0 or higher dataset standards)

#### **Generation of Rich Text Format (RTF) Files**

• RTF files will be generated for summary displays.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.

#### **Reporting Standards**

• The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - o Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - o Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| <b>Descriptive Summary</b> | Descriptive Summary Statistics |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary<br>Statistics | Refer to IDSL Statistical Principle 6.06.1 Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharmac | cokinetic Parameters |
| Descriptive Summary Statistics. (Un-Transformed) | N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum and CV(%) • CV(%)=(SD/mean)*100 |
| Descriptive Summary Statistics. (Log <sub>e</sub> Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between-subject geometric coefficient of variation (CV<sub>b</sub> (%)) will be reported.</li> <li>Geometric mean = exp (mean on log<sub>e</sub> scale)</li> <li>CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 [NOTE: SD = SD of log<sub>e</sub> transformed data]</li> </ul> |
| Parameters Not Being Loge Transformed | $\%$ AUC <sub>ex</sub> , $T_{max}$ , $t_{lag}$ , $t$ , $\lambda z$ , $Vz/F$ |
| Listings | Include PK Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , % $AUC_{ex}$ , $C_{max}$ , $C_{24}$ , $C_{t}$ , $C_{t}$ , $C_{max}$ , $C_{24}$ , $C_{t}$ , $C_{t$ |

#### CONFIDENTIAL

| Reporting Standards | |
|---|---|
| | reference) for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{24}$ and $C_{max}$ ; and the ratio of $AUC_{(0-t)}/AUC_{(0-\infty)}$ ( $AUC_t(\%)$ ) for Canada specific submission requirement. |
| Graphical Displays | |
| • Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. **General**

# **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.

#### **Study Day**

- Calculated as the number of days from Treatment start date :
  - Ref Date = Missing  $\rightarrow$  Study Day = Missing
  - Ref Date < Treatment start Date → Study Day = Ref Date Treatment start Date
  - Ref Data ≥ Treatment start Date → Study Day = (Ref Date Treatment start Date) + 1

# 10.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age using date of the screening visit relative to birth date, where birth date is imputed as:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

# 10.6.3. Safety

#### **ECG Parameters**

#### **RR** Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as :

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = [(QT/QTcB)^{(2)}]*1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = [(QT/QTcF)^{(3)}]*1000$$

#### **Corrected QT Intervals**

• When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

• IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

• Example 1: 2 Significant Digits = '< x' becomes x - 0.01

• Example 2: 1 Significant Digit = '> x' becomes x + 0.1

• Example 3: 0 Significant Digits = '< x' becomes x – 1

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>All subjects who withdraw prematurely from the study/study drug will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR).</li> <li>All available data collected up until the point of withdrawal, and the follow-up visits will be used in the analyses and will be listed and all available planned data will be included in the summaries according to the populations defined in Section 4.</li> <li>Any data collected up until the point of withdrawal, and the follow-up visits will be used in the analyses.</li> <li>In the event that the study is prematurely discontinued, all available data will be listed and a review carried out by the study team to assess which statistical analyses are still considered appropriate.</li> </ul> |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |

# 10.7.2.2. Handling of PK Concentration Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>The PK Plasma Concentration Population will include all subjects who undergo plasma PK sampling and have evaluable PK assay results for DTG or 3TC.</li> <li>Data from subjects who vomit within 4 hours of study drug administration or who have major protocol deviations will be excluded from PK concentration summary, PK parameter summary and statistical comparisons but will be included in the Listing and flagged.</li> <li>This population will be used for listing PK concentrations, parameters, calculating PK parameters and plotting of individual concentration-time files.</li> <li>If the pre-dose concentration is ≤ 5% of Cmax value in a subject, the concentration data for that subject without any adjustments will be included in PK and statistical analysis. If the pre-dose concentration is &gt; 5% of Cmax value in a subject, then the concentration data for that subject will not be included in PK and statistical analysis and only the concentration data of that subject(s) will be presented</li> <li>If during clinical phase, 3 consecutive samples in any phase i.e. (Absorption, Distribution and Metabolism / Excretion) are found to be missing then data for that subject will not be included in PK and statistical analysis and only the concentration data of that subject(s) will be presented</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

Division of AIDS (DAIDS, Version 2.0, November 2014) AE grade 2 and above of lab abnormalities will be listed by subject, period/treatment, visit, and actual date and time.

#### 10.8.2. ECG

# **ECG Values of Potential Clinical Importance (Healthy Volunteers)**

| ECG Parameter | Potential Clinical Importance Range (PCI) | Unit |
|-----------------------|-------------------------------------------|------|
| Absolute QTc Interval | >450 | msec |
| PR Interval | <110 and >220 | msec |
| QRS Interval | <75 and >110 | msec |

# 10.8.3. Vital Signs

#### **Vital Signs Values of Potential Clinical Importance (Healthy Volunteers)**

| VS Parameter | Potential Clinical Importance Range (PCI) | Unit |
|--------------------------|-------------------------------------------|------|
| Systolic Blood Pressure | <85 and >160 | mmHg |
| Diastolic Blood Pressure | <45 and >100 | mmHg |
| Heart Rate | <40 and >110 | bpm |

#### Vital Signs change from Baseline Flagging Range

| VS Parameter | Flagging Criteria | Unit |
|--------------------------|--------------------|------|
| Systolic Blood Pressure | Increase ≥20 | mmHg |
| (Change from Baseline) | Increase ≥40 | |
| | Decrease ≥ 20 | |
| | Decrease≥40 | |
| Diastolic Blood Pressure | Increase $\geq 10$ | mmHg |
| (Change from Baseline) | Increase≥20 | |
| | Decrease ≥ 10 | |
| | Decrease≥20 | |
| Heart Rate | Increase ≥ 15 | bpm |
| (Change from Baseline) | Increase ≥ 30 | |
| | Decrease ≥ 15 | ] |
| | Decrease ≥ 30 | ] |

# 10.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

#### 10.9.1. Statistical Analysis Assumptions

| Endpoint(s) | • AUC(0-∞), AUC(0-t), Cmax, CL/F, AUC(0-24), C24, t1/2 |
|-------------|--------------------------------------------------------|
| Analysis | Linear Mixed Model |

#### **Assumptions:**

- For the Linear Mixed Model, model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the G matrix will be used by specifying 'type=UN' on the RANDOM line.
  - o In the event that this model fails to converge, alternative covariance structures may be considered such as VC or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- Sensitivity analysis will be performed if the normality assumptions are violated due to presence of outliers.

# 10.10. Appendix 10 - Abbreviations & Trade Marks

# 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| ADaM IG | Analysis Data Model Implementation Guide |
| AE | Adverse Event |
| AUC | Area under concentration-time curve |
| $AUC_{(0-\infty)}$ | Area under the concentration-time curve from time zero (pre-dose) |
| , | extrapolated to infinite time |
| AUC <sub>(0-t)</sub> | Area under the concentration-time curve from time zero (pre-dose) to |
| | last time of quantifiable concentration |
| $AUC_{(0-24)}$ | Area under the plasma concentration time curve from time zero to 24 |
| | hours |
| %AUC <sub>ex</sub> | % of AUC( $0-\infty$ ) that was extrapolated |
| $AUC_t(\%)$ | Percent of the area measured by AUC(0-t) relative to the extrapolated |
| | $AUC(0-\infty)$ |
| BE | Bioequivalence |
| BESM | Bioanalytical External Study Monitors |
| BIB | Bioanalysis, Immunogenicity and Biomarkers |
| $C_{24}$ | Drug concentration at 24 hours post-dose |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | The apparent oral clearance |
| $C_{max}$ | Maximum observed concentration |
| CP | Clinical Programming |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSSO | Clinical Pharmacology Sciences and Study Operations |
| CRF | Case record form |
| CS | Clinical Statistics |
| $C_{t}$ | last quantifiable concentration |
| CV | Coefficient of Variation |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between)/Coefficient of Variation (Within) |
| DAIDS | Division of Acquired Immune Deficiency Syndrome |
| DBF | Database Freeze |
| DBR | Database Release |
| DTG | Dolutegravir |
| FD | Food Effect |
| GSK | GlaxoSmithKline |
| HARP | Harmonized Analysis and Reporting Process |
| IDSL | Integrated Data Standards Library |
| λz | Terminal phase rate constant |
| LLQ | Lower limit of quantification |
| NC | Not Calculable |

| NQ | Non-quantifiable concentration measured as below LLQ |
|------------------|------------------------------------------------------|
| PK | Pharmacokinetic |
| QSci | Quantitative Sciences |
| RAP | Reporting and Analysis Plan |
| RTF | Rich Text Format |
| 3TC | Lamivudine, EPIVIR <sup>TM</sup> |
| SAS | Statistical Analysis System |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SRP | Statistics Resourcing and Programming |
| t | time of last quantifiable concentration |
| t <sub>1/2</sub> | Terminal phase half-life |
| $t_{lag}$ | Absorption lag time |
| $T_{max}$ | Time of occurrence of Cmax |
| $\lambda z$ | Apparent elimination rate constant |
| Vz/F | Apparent oral volume of distribution |

# 10.10.2. Trademarks

| Trademarks of ViiV Healthcare |
|-------------------------------|
| EPIVIR |
| EPZICOM |
| TIVICAY |
| TRIUMEQ |
| TRIZIVIR |

| Trademarks not owned by ViiV<br>Healthcare |
|--------------------------------------------|
| MedDRA |
| SAS |
| WinNonlin |
## 10.11. Appendix 11: List of Data Displays

### 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|---|---|---|
| Study Population | 1.01 to 1.05 | N/A |
| Pharmacokinetic | 2.01 to 2.78* | 2.01 to 2.44* |
| | *If Part 2 is conducted, same set | *If Part 2 is conducted, same set |
| | of tables will be provided as | of figures will be provided as |
| | 2.101 to 2.178 with Part 1 and | 2.101 to 2.144 with Part 1 and |
| | Part 2 indication in the titles | Part 2 indication in the titles |
| Safety | 3.01 to 3.13* | N/A |
| | *If Part 2 is conducted, same set | |
| | of tables will be provided as | |
| | 3.101 to 3.113 with Part 1 and | |
| | Part 2 indication in the titles | |
| Section | List | ings* |
| | *If Part 2 is conducted, same set of | of listings will be provided as 101 |
| | to 148 with Part 1 and Part 2 indication in the titles | |
| ICH Listings | 1 to 25 | |
| Other Listings | 26 1 | to 48 |

## 10.11.2. Mock Example Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------------|---------------------|---------|
| Study Population | N/A | N/A | N/A |
| Pharmacokinetic | PK_F1, PK_F2 | PK_T1, PK_T2, | N/A |
| | | PK_T3, PK_T4, PK_T5 | |
| Safety | N/A | SAFE_T1 | SAFE_L1 |

#### **NOTES:**

• Indicate display is Non-Standard in the 'IDSL/TST ID / Example Shell' or 'Programming Notes' column.

# 10.11.3. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | et Disposition | | | | |
| 1.01 | Safety | CP_ES1 (XO) | Summary of Subject Disposition | Include Part 2 and Total (if Part 2 is conducted) | SAC |
| Demog | graphics | | | | |
| 1.02 | Safety | DM3 (XO) | Summary of Demographic characteristics | Include BMI, Race detail<br>Include Part 2 and Total (if Part 2 is<br>conducted) | SAC |
| 1.03 | Safety | DM5 | Summary of Race and Racial<br>Combinations | Include Part 2 and Total (if Part 2 is conducted) | SAC |
| 1.04 | Safety | DM6 | Summary of Race and Racial<br>Combinations Details | Include Part 2 and Total (if Part 2 is conducted) | SAC |
| 1.05 | Safety | DV1 | Summary of Important Protocol<br>Deviations | Include Part 2 and Total (if Part 2 is conducted) | SAC |

### 10.11.4. Pharmacokinetic Tables

## If Part 2 is conducted, same set of tables will be provided as 2.101 to 2.178 with Part 1 and Part 2 indication in the titles

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| PK Co | ncentration Data | | | | |
| 2.01 | PK Parameter<br>BE Summary | pkct1 | Summary of DTG Plasma Concentration-time<br>Data (unit) by Treatment - Bioequivalence<br>Assessment | Treatments A, B only | SAC |
| 2.02 | PK Parameter<br>BE Summary | pkct1 | Summary of 3TC Plasma Concentration-time Data (unit) by Treatment - Bioequivalence Assessment | Treatments A, B only | SAC |
| 2.03 | PK Parameter<br>FD Summary | pkct1 | Summary of DTG Plasma Concentration-time Data (unit) by Treatment - Food Effect | Treatments B, B_Fed only | SAC |
| 2.04 | PK Parameter<br>FD Summary | pkct1 | Summary of 3TC Plasma Concentration-time Data (unit) by Treatment – Food Effect | Treatments B, B_Fed only | SAC |
| 2.05 | PK Plasma<br>Concentration | pkct1 | Summary of DTG Plasma Concentration-time<br>Data (unit) by Treatment | All 3 treatments in the same table | SAC |
| 2.06 | PK Plasma<br>Concentration | pkct1 | Summary of 3TC Plasma Concentration-time Data (unit) by Treatment | All 3 treatments in the same table | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK De | rived Parameters | based on Actual S | Sampling Time | | |
| 2.07 | PK Parameter<br>BE Summary | pkpt1 | Summary of Untransformed DTG Plasma PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.08 | PK Parameter<br>BE Summary | pkpt1 | Summary of Untransformed 3TC Plasma PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.09 | PK Parameter<br>BE Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed DTG Plasma PK<br>Parameters based on Actual Sampling Time -<br>Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units;<br>Treatments A, B only | SAC |
| 2.10 | PK Parameter<br>BE Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK<br>Parameters based on Actual Sampling Time -<br>Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units;<br>Treatments A, B only | SAC |
| 2.11 | PK Parameter<br>FD Summary | pkpt1 | Summary of Untransformed DTG Plasma PK Parameters based on Actual Sampling Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |
| 2.12 | PK Parameter<br>FD Summary | pkpt1 | Summary of Untransformed 3TC Plasma PK Parameters based on Actual Sampling Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13 | PK Parameter<br>FD Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed DTG Plasma PK<br>Parameters based on Actual Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units;<br>Treatments B, B Fed only | SAC |
| 2.14 | PK Parameter<br>FD Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK<br>Parameters based on Actual Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.15 | PK Plasma<br>Concentration | pkpt1 | Summary of Untransformed DTG Plasma PK<br>Parameters based<br>on Actual Sampling Time | All parameters with units;<br>All treatments | SAC |
| 2.16 | PK Plasma<br>Concentration | pkpt1 | Summary of Untransformed 3TC Plasma PK<br>Parameters based<br>on Actual Sampling Time | All parameters with units;<br>All treatments | SAC |
| 2.17 | PK Plasma<br>Concentration | pkpt3 | Summary of Log <sub>e</sub> -transformed DTG Plasma PK<br>Parameters based on Actual Sampling Time | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units;<br>All treatments | SAC |
| 2.18 | PK Plasma<br>Concentration | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK Parameters based on Actual Sampling Time | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with units; All treatments | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Statist | ical Analysis Table | e based on Actual | | | |
| 2.19 | PK Parameter<br>BE Summary | PK_T1 | Summary of Statistical Analysis of Loge-<br>transformed DTG Plasma PK Parameters based<br>on Actual Sampling Time - Bioequivalence<br>Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $CL/F$ and $t_{1/2}$ with<br>units; Treatments A, B only | SAC |
| 2.20 | PK Parameter<br>BE Summary | PK_T1 | Summary of Statistical Analysis of Loge-<br>transformed 3TC Plasma PK Parameters based on<br>Actual Sampling Time - Bioequivalence<br>Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $CL/F$ and $t_{1/2}$ with<br>units; Treatments A, B only | SAC |
| 2.21 | PK Parameter<br>BE Summary | PK_T2 | Summary of Statistical Analysis of<br>Untransformed DTG Plasma PK Parameters<br>based on Actual Sampling Time - Bioequivalence<br>Assessment | Parameters $t_{lag}$ and $T_{max}$ with units; Treatments A, B only | SAC |
| 2.22 | PK Parameter<br>BE Summary | PK_T2 | Summary of Statistical Analysis of Untransformed 3TC Plasma PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | Parameters $t_{lag}$ and $T_{max}$ with units; Treatments A, B only | SAC |
| 2.23 | PK Parameter<br>BE Summary | MID201676,<br>Table 2.17 | Summary of Type 3 Tests of Fixed Effects for Loge-transformed PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.24 | PK Parameter<br>BE Summary | MID201676,<br>Table 2.18 | Summary of Variance Estimates Effects for PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.25 | PK Parameter<br>FD Summary | PK_T1 | Summary of Statistical Analysis of Loge-<br>transformed DTG Plasma PK Parameters based<br>on Actual Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.26 | PK Parameter<br>FD Summary | PK_T1 | Summary of Statistical Analysis of Logetransformed 3TC Plasma PK Parameters based on Actual Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.27 | PK Parameter<br>FD Summary | PK_T2 | Summary of Statistical Analysis of Untransformed DTG Plasma PK Parameters based on Actual Sampling Time – Food Effect | Parameters t <sub>lag</sub> and T <sub>max</sub> with units; Treatments B, B Fed only | SAC |
| 2.28 | PK Parameter<br>FD Summary | PK_T2 | Summary of Statistical Analysis of Untransformed 3TC Plasma PK Parameters based on Actual Sampling Time – Food Effect | Parameters t <sub>lag</sub> and T <sub>max</sub> with units; Treatments B, B_Fed only | SAC |
| 2.29 | PK Parameter<br>FD Summary | MID201676,<br>Table 2.17 | Summary of Type 3 Tests of Fixed Effects for Loge-transformed PK Parameters based on Actual Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.30 | PK Parameter<br>FD Summary | MID201676,<br>Table 2.18 | Summary of Variance Estimates Effects for PK<br>Parameters based on Actual Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| PK De | rived Parameters | based on Nomina | | | |
| 2.31 | PK Parameter<br>BE Summary | pkpt1 | Summary of Untransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.32 | PK Parameter<br>BE Summary | pkpt1 | Summary of Untransformed 3TC Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.33 | PK Parameter<br>BE Summary | pkpt3 | Summary of Loge-transformed DTG Plasma PK<br>Parameters based on Nominal Sampling Time -<br>Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units; Treatments A, B only | SAC |
| 2.34 | PK Parameter<br>BE Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK<br>Parameters based on Nominal Sampling Time -<br>Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units; Treatments A, B only | SAC |
| 2.35 | PK Parameter<br>FD Summary | pkpt1 | Summary of Untransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |
| 2.36 | PK Parameter<br>FD Summary | pkpt1 | Summary of Untransformed 3TC Plasma PK Parameters based on Nominal Sampling Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |
| 2.37 | PK Parameter<br>FD Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed DTG Plasma PK<br>Parameters based on Nominal Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.38 | PK Parameter<br>FD Summary | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK<br>Parameters based on Nominal Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.39 | PK Plasma<br>Concentration | pkpt1 | Summary of Untransformed DTG Plasma PK Parameters based on Nominal Sampling Time | All parameters with units;<br>All treatments | SAC |
| 2.40 | PK Plasma<br>Concentration | pkpt1 | Summary of Untransformed 3TC Plasma PK<br>Parameters based on Nominal Sampling Time | All parameters with units;<br>All treatments | SAC |
| 2.41 | PK Plasma<br>Concentration | pkpt3 | Summary of Log <sub>e</sub> -transformed DTG Plasma PK Parameters based on Nominal Sampling Time | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units; All treatments | SAC |
| 2.42 | PK Plasma<br>Concentration | pkpt3 | Summary of Log <sub>e</sub> -transformed 3TC Plasma PK<br>Parameters based on Nominal Sampling Time | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $C_t$ , $CL/F$ and $t_{1/2}$ with<br>units; All treatments | SAC |
| Statist | ical Analysis Table | e based on Nomin | al Sampling Time | | |
| 2.43 | PK Parameter<br>BE Summary | PK_T1 | Summary of Statistical Analysis of Logetransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | $ \begin{array}{c} \text{IA (only} \\ \text{AUC}_{(0\text{-}\infty)}, \\ \text{AUC}_{(0\text{-}t)}, \\ \text{C}_{\text{max}}) \\ \text{SAC} \end{array} $ |

| Pharm | nacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.44 | PK Parameter<br>BE Summary | PK_T1 | Summary of Statistical Analysis of Logetransformed 3TC Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | $\begin{array}{c} \text{IA (only} \\ \text{AUC}_{(0\text{-}\infty)}, \\ \text{AUC}_{(0\text{-}t)}, \\ \text{C}_{\text{max}}) \\ \text{SAC} \end{array}$ |
| 2.45 | PK Parameter<br>BE Summary | PK_T2 | Summary of Statistical Analysis of Untransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Parameters tlag and Tmax with units; Treatments A, B only | SAC |
| 2.46 | PK Parameter<br>BE Summary | PK_T2 | Summary of Statistical Analysis of<br>Untransformed 3TC Plasma PK Parameters based<br>on Nominal Sampling Time - Bioequivalence<br>Assessment | Parameters tlag and Tmax with units; Treatments A, B only | SAC |
| 2.47 | PK Parameter<br>BE Summary | MID201676,<br>Table 2.17 | Summary of Type 3 Tests of Fixed Effects for Loge-transformed PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.48 | PK Parameter<br>BE Summary | MID201676,<br>Table 2.18 | Summary of Variance Estimates Effects for PK<br>Parameters based on Nominal Sampling Time -<br>Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ ,<br>$AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ ,<br>$C_{24}$ , $CL/F$ and $t_{1/2}$ with<br>units; Treatments A, B only | SAC |
| 2.49 | PK Parameter<br>FD Summary | PK_T1 | Summary of Statistical Analysis of Loge-<br>transformed DTG Plasma PK Parameters based<br>on Nominal Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | $\begin{array}{c} \text{IA (only} \\ \text{AUC}_{(0\text{-}\infty)}, \\ \text{AUC}_{(0\text{-}t)}, \\ \text{C}_{\text{max}}) \\ \text{SAC} \end{array}$ |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.50 | PK Parameter<br>FD Summary | PK_T1 | Summary of Statistical Analysis of Loge-<br>transformed 3TC Plasma PK Parameters based on<br>Nominal Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | IA (only $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $C_{max}$ ) SAC |
| 2.51 | PK Parameter<br>FD Summary | PK_T2 | Summary of Statistical Analysis of Untransformed DTG Plasma PK Parameters based on Nominal Sampling Time – Food Effect | Parameters t <sub>lag</sub> and T <sub>max</sub> with units; Treatments B, B_Fed only | SAC |
| 2.52 | PK Parameter<br>FD Summary | PK_T2 | Summary of Statistical Analysis of<br>Untransformed 3TC Plasma PK Parameters based<br>on Nominal Sampling Time – Food Effect | Parameters t <sub>lag</sub> and T <sub>max</sub> with units; Treatments B, B_Fed only | SAC |
| 2.53 | PK Parameter<br>FD Summary | ING114580,<br>Table 3.10 | Summary of Type 3 Tests of Fixed Effects for Log <sub>e</sub> -transformed PK Parameters based on Nominal Sampling Time - Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.54 | PK Parameter<br>FD Summary | ING114580,<br>Table 3.11 | Summary of Variance Estimates Effects for PK<br>Parameters based on Nominal Sampling Time -<br>Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| | Canada Specific PK Tables | | | | |
| PK Co | PK Concentration Data | | | | |
| 2.55 | PK Plasma<br>Concentration | PK_T3 | DTG Drug Concentration (unit) for the Test<br>Formulation B | | SAC |

| Pharm | nacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| 2.56 | PK Plasma<br>Concentration | PK_T3 | DTG Drug Concentration (unit) for the Test<br>Formulation B_Fed | | SAC |
| 2.57 | PK Plasma<br>Concentration | PK_T3 | DTG Drug Concentration (unit) for the Reference Formulation A | | SAC |
| 2.58 | PK Plasma<br>Concentration | PK_T3 | 3TC Drug Concentration (unit) for the Test<br>Formulation B | | SAC |
| 2.59 | PK Plasma<br>Concentration | PK_T3 | 3TC Drug Concentration (unit) for the Test Formulation B_Fed | | SAC |
| 2.60 | PK Plasma<br>Concentration | PK_T3 | 3TC Drug Concentration (unit) for the Reference Formulation A | | SAC |
| PK De | rived Parameters | based on Actual S | Sampling Time | | • |
| 2.61 | PK Plasma<br>Concentration | PK_T4 | DTG Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B | All parameters with units | SAC |
| 2.62 | PK Plasma<br>Concentration | PK_T4 | DTG Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B_Fed | All parameters with units | SAC |
| 2.63 | PK Plasma<br>Concentration | PK_T4 | DTG Parameter Estimates based on Actual Time for Each Subject Given the Reference Formulation A | All parameters with units | SAC |
| 2.64 | PK Plasma<br>Concentration | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B | All parameters with units | SAC |
| 2.65 | PK Plasma<br>Concentration | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B_Fed | All parameters with units | SAC |
| 2.66 | PK Plasma<br>Concentration | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Reference Formulation A | All parameters with units | SAC |

| Pharn | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.67 | PK Parameter<br>BE Summary | PK_T4 | DTG Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B - Bioequivalence Assessment | All parameters with units | SAC |
| 2.68 | PK Parameter<br>BE Summary | PK_T4 | DTG Parameter Estimates based on Actual Time<br>for Each Subject Given the Reference<br>Formulation A - Bioequivalence Assessment | All parameters with units | SAC |
| 2.69 | PK Parameter<br>BE Summary | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B - Bioequivalence Assessment | All parameters with units | SAC |
| 2.70 | PK Parameter<br>BE Summary | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Reference Formulation A - Bioequivalence Assessment | All parameters with units | SAC |
| 2.71 | PK Parameter<br>BE Summary | PK_T5 | DTG Parameter Analysis – Data based on Actual<br>Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.72 | PK Parameter<br>BE Summary | PK_T5 | 3TC Parameter Analysis – Data based on Actual<br>Time - Bioequivalence Assessment | All parameters with units;<br>Treatments A, B only | SAC |
| 2.73 | PK Parameter<br>FD Summary | PK_T4 | DTG Parameter Estimates based on Actual Time for Each Subject Given the Test Formulation B Fed – Food Effect | All parameters with units | SAC |
| 2.74 | PK Parameter<br>FD Summary | PK_T4 | DTG Parameter Estimates based on Actual Time<br>for Each Subject Given the Reference<br>Formulation A – Food Effect | All parameters with units | SAC |
| 2.75 | PK Parameter<br>FD Summary | PK_T4 | 3TC Parameter Estimates based on Actual Time<br>for Each Subject Given the Test Formulation<br>B_Fed – Food Effect | All parameters with units | SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.76 | PK Parameter<br>FD Summary | PK_T4 | 3TC Parameter Estimates based on Actual Time for Each Subject Given the Reference Formulation A – Food Effect | All parameters with units | SAC |
| 2.77 | PK Parameter<br>FD Summary | PK_T5 | DTG Parameter Analysis – Data based on Actual<br>Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |
| 2.78 | PK Parameter<br>FD Summary | PK_T5 | 3TC Parameter Analysis – Data based on Actual Time - Food Effect | All parameters with units;<br>Treatments B, B_Fed only | SAC |

## 10.11.5. Pharmacokinetic Figures

## If Part 2 is conducted, same set of figures will be provided as 2.101 to 2.144 with Part 1 and Part 2 indication in the titles

| Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Indivi | dual Concentratio | on Plots | | | |
| 2.01 | PK Plasma<br>Concentration | pkcflx | Individual Subject DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) by Subject | Paged by Subject | SAC |
| 2.02 | PK Plasma<br>Concentration | pkcflx | Individual Subject 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) by Subject | Paged by Subject | SAC |
| 2.03 | PK Plasma<br>Concentration | pkcf6 | Individual Subject DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) by Treatment | Paged by Treatment | SAC |
| 2.04 | PK Plasma<br>Concentration | pkcf6 | Individual Subject 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) by Treatment | Paged by Treatment | SAC |

| Pharn | nacokinetic Figur | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Mean | / Median Concen | tration Plots | | | |
| 2.05 | PK Parameter<br>BE Summary | pkcf4 | Arithmetic Mean (+SD) DTG Plasma<br>Concentration-time Plot (Linear and Semi-log)<br>- Bioequivalence Assessment | Use nominal times in X Axis, Paged by Treatment. Treatments A, B only | SAC |
| 2.06 | PK Parameter<br>BE Summary | pkcf4 | Arithmetic Mean (+SD) 3TC Plasma<br>Concentration-time Plot (Linear and Semi-log)<br>- Bioequivalence Assessment | Use nominal times in X Axis, Paged by Treatment. Treatments A, B only | SAC |
| 2.07 | PK Parameter<br>BE Summary | pkcf5 | Median (range) DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) -<br>Bioequivalence Assessment | Use nominal times in X Axis, Paged by Treatment. Treatments A, B only | SAC |
| 2.08 | PK Parameter<br>BE Summary | pkcf5 | Median (range) 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) -<br>Bioequivalence Assessment | Use nominal times in X Axis, Paged by Treatment. Treatments A, B only | SAC |
| 2.09 | PK Parameter<br>BE Summary | pkcf4 | Arithmetic Mean DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) -<br>Bioequivalence Assessment | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments A, B only | SAC |
| 2.10 | PK Parameter<br>BE Summary | pkcf4 | Arithmetic Mean 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) -<br>Bioequivalence Assessment | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments A, B only | SAC |

| Pharn | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11 | PK Parameter<br>BE Summary | pkcf5 | Median DTG Plasma Concentration-time Plot<br>(Linear and Semi-log) - Bioequivalence<br>Assessment | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments A, B only | SAC |
| 2.12 | PK Parameter<br>BE Summary | pkcf5 | Median 3TC Plasma Concentration-time Plot<br>(Linear and Semi-log)- Bioequivalence<br>Assessment | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments A, B only | SAC |
| 2.13 | PK Parameter<br>FD Summary | pkcf4 | Arithmetic Mean (+SD) DTG Plasma<br>Concentration-time Plot (Linear and Semi-log)<br>- Food Effect | Use nominal times in X Axis, Paged by Treatment. Treatments B, B_Fed only | SAC |
| 2.14 | PK Parameter<br>FD Summary | pkcf4 | Arithmetic Mean (+SD) 3TC Plasma Concentration-time Plot (Linear and Semi-log) - Food Effect | Use nominal times in X Axis, Paged by Treatment. Treatments B, B_Fed only | SAC |
| 2.15 | PK Parameter<br>FD Summary | pkcf5 | Median (range) DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) - Food Effect | Use nominal times in X Axis, Paged by Treatment. Treatments B, B_Fed only | SAC |
| 2.16 | PK Parameter<br>FD Summary | pkcf5 | Median (range) 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) - Food Effect | Use nominal times in X Axis, Paged by Treatment. Treatments B, B_Fed only | SAC |

| Pharn | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.17 | PK Parameter<br>FD Summary | pkcf4 | Arithmetic Mean DTG Plasma Concentration-<br>time Plot (Linear and Semi-log) - Food Effect | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments B, B Fed only | SAC |
| 2.18 | PK Parameter<br>FD Summary | pkcf4 | Arithmetic Mean 3TC Plasma Concentration-<br>time Plot (Linear and Semi-log) - Food Effect | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments B, B Fed only | SAC |
| 2.19 | PK Parameter<br>FD Summary | pkcf5 | Median DTG Plasma Concentration-time Plot<br>(Linear and Semi-log) - Food Effect | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments B, B Fed only | SAC |
| 2.20 | PK Parameter<br>FD Summary | pkcf5 | Median 3TC Plasma Concentration-time Plot<br>(Linear and Semi-log) - Food Effect | Use nominal times in X Axis. Keep all the treatments in one plot. Use different colours for different treatments. Treatments B, B_Fed only | SAC |
| Comp | arative PK Paran | neters Plots bas | sed on Actual Sampling Time | | |
| 2.21 | PK Parameter<br>BE Summary | pkpf3 | Comparative Plot of Individual Subject DTG Plasma Pharmacokinetic Parameter based on Actual Sampling Time Versus Treatment - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |

| Pharm | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.22 | PK Parameter<br>BE Summary | pkpf3 | Comparative Plot of Individual Subject 3TC Plasma Pharmacokinetic Parameter based on Actual Sampling Time Versus Treatment - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.23 | PK Parameter<br>BE Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects DTG Plasma Pharmacokinetic<br>Parameters based on Actual Sampling Time -<br>Bioequivalence Assessment | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.24 | PK Parameter<br>BE Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects 3TC Plasma Pharmacokinetic<br>Parameters based on Actual Sampling Time -<br>Bioequivalence Assessment | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.25 | PK Parameter<br>FD Summary | pkpf3 | Comparative Plot of Individual Subject DTG Plasma Pharmacokinetic Parameter based on Actual Sampling Time Versus Treatment – Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.26 | PK Parameter<br>FD Summary | pkpf3 | Comparative Plot of Individual Subject 3TC Plasma Pharmacokinetic Parameter based on Actual Sampling Time Versus Treatment – Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |

| Pharm | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27 | PK Parameter<br>FD Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects DTG Plasma Pharmacokinetic<br>Parameters based on Actual Sampling Time –<br>Food Effect | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.28 | PK Parameter<br>FD Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects 3TC Plasma Pharmacokinetic<br>Parameters based on Actual Sampling Time –<br>Food Effect | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| Statist | ical Analysis Plot | s based on Act | ual Sampling Time | | |
| 2.29 | PK Parameter<br>BE Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of DTG Plasma Pharmacokinetic Parameters based on Actual Sampling Time - Bioequivalence Assessment | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments A, B only | SAC |
| 2.30 | PK Parameter<br>BE Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of 3TC Plasma Pharmacokinetic Parameters based on Actual Sampling Time - Bioequivalence Assessment | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments A, B only | SAC |
| 2.31 | PK Parameter<br>FD Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of DTG Plasma Pharmacokinetic Parameters based on Actual Sampling Time – Food Effect | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments B, B_Fed only | SAC |

| Pharn | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.32 | PK Parameter<br>FD Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of 3TC Plasma Pharmacokinetic Parameters based on Actual Sampling Time – Food Effect | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments B, B_Fed only | SAC |
| Comp | arative PK Paran | neters Plots ba | sed on Nominal Sampling Time | | 1 |
| 2.33 | PK Parameter<br>BE Summary | pkpf3 | Comparative Plot of Individual Subject DTG Plasma Pharmacokinetic Parameter based on Nominal Sampling Time Versus Treatment - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.34 | PK Parameter<br>BE Summary | pkpf3 | Comparative Plot of Individual Subject 3TC Plasma Pharmacokinetic Parameter based on Nominal Sampling Time Versus Treatment - Bioequivalence Assessment | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.35 | PK Parameter<br>BE Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects DTG Plasma Pharmacokinetic<br>Parameters based on Nominal Sampling Time -<br>Bioequivalence Assessment | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |
| 2.36 | PK Parameter<br>BE Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects 3TC Plasma Pharmacokinetic<br>Parameters based on Nominal Sampling Time -<br>Bioequivalence Assessment | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments A, B only | SAC |

| Pharm | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.37 | PK Parameter<br>FD Summary | pkpf3 | Comparative Plot of Individual Subject DTG Plasma Pharmacokinetic Parameter based on Nominal Sampling Time Versus Treatment – Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.38 | PK Parameter<br>FD Summary | pkpf3 | Comparative Plot of Individual Subject 3TC Plasma Pharmacokinetic Parameter based on Nominal Sampling Time Versus Treatment – Food Effect | Parameters $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.39 | PK Parameter<br>FD Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects DTG Plasma Pharmacokinetic<br>Parameters based on Nominal Sampling Time –<br>Food Effect | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| 2.40 | PK Parameter<br>FD Summary | PK_F1 | Treatment Comparative Plot of Adjusted<br>Geometric Mean (95% CI) with Individual<br>Subjects 3TC Plasma Pharmacokinetic<br>Parameters based on Nominal Sampling Time –<br>Food Effect | Paged by $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ with units; Treatments B, B_Fed only | SAC |
| Statist | ical Analysis Plot | s based on Nor | ninal Sampling Time | | |
| 2.41 | PK Parameter<br>BE Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of DTG Plasma Pharmacokinetic Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments A, B only | SAC |

| Pharm | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.42 | PK Parameter<br>BE Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of 3TC Plasma Pharmacokinetic Parameters based on Nominal Sampling Time - Bioequivalence Assessment | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments A, B only | SAC |
| 2.43 | PK Parameter<br>FD Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of DTG Plasma Pharmacokinetic Parameters based on Nominal Sampling Time – Food Effect | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments B, B_Fed only | SAC |
| 2.44 | PK Parameter<br>FD Summary | PK_F2 | Geometric Mean Treatment Ratio and 90% CI of 3TC Plasma Pharmacokinetic Parameters based on Nominal Sampling Time – Food Effect | Produce for $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $AUC_{(0-24)}$ , $C_{max}$ , $C_{24}$ , $CL/F$ and $t_{1/2}$ , all parameters on one plot. Treatments B, B_Fed only | SAC |

## 10.11.6. Safety Tables

## If Part 2 is conducted, same set of tables will be provided as 3.101 to 3.113 with Part 1 and Part 2 indication in the titles

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| Adver | rse Events | | | | |
| 3.01 | Safety | CP_AE1x (xo) | Summary of All Adverse Events | | SAC |
| 3.02 | Safety | CP_AE1x (xo) | Summary of Drug-Related Adverse Events | | SAC |
| 3.03 | Safety | CP_AE1x (xo) | Summary of Serious Adverse Events | | SAC |
| 3.04 | Safety | CP_AE1x (xo) | Summary of AEs Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | SAC |
| Labs | | • | | | |
| 3.05 | Safety | LB1 | Summary of Chemistry Laboratory Values | | SAC |
| 3.06 | Safety | LB1 | Summary of Change from Baseline for<br>Chemistry Laboratory Values | | SAC |
| 3.07 | Safety | LB1 | Summary of Hematology Laboratory Values | | SAC |
| 3.08 | Safety | LB1 | Summary of Change from Baseline for<br>Hematology Laboratory Values | | SAC |
| <b>ECGs</b> | | | | | |
| 3.09 | Safety | EG1 | Summary of ECG Findings | | SAC |
| 3.10 | Safety | EG2 | Summary of ECG Values | | SAC |
| Vital S | Signs | | | | |
| 3.11 | Safety | VS1 | Summary of Vital Signs | Include BP, HR | SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12 | Safety | VS1 | Summary of Change From Baseline for Vital<br>Signs | Include BP, HR | SAC |
| 3.13 | Safety | SAFE_T1 | Frequency of Subjects with Vital Signs Measurements Outside the Potential Clinical Concern Range | | SAC |

# **10.11.7. ICH Listings**

## If Part 2 is conducted, same set of listings will be provided as 101 to 148 with Part 1 and Part 2 indication in the titles

| ICH | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Ran | domisation | | | | |
| 1 | Safety | CP_RA1x (XO) | Listing of Randomized and Actual Treatments | Add randomization date | SAC |
| Subj | ect Disposition | | | | |
| 2 | Screening | ES7 | Listing of Reasons for Screening Failures | Include Age and Sex. Concatenate with Subjid | SAC |
| 3 | Safety | CP_ES10x<br>(XO) | Listing of Reasons for Withdrawal | | SAC |
| 4 | Safety | DV2 | Listing of Protocol Deviations | | SAC |
| 5 | Screening | SAFE_L1 | Listing of Subjects Excluded from<br>Analysis Populations | | SAC |
| 6 | Safety | IE4 (XO) | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Dem | ographics | | | | |
| 7 | Safety | DM4 (XO) | Listing of Demographic Characteristics | | SAC |
| 8 | Safety | DM10 (XO) | Listing of Race | | SAC |
| Concomitant Medication | | | | | |
| 9 | Safety CP_CM4 Listing of Concomitant Medications by Generic Term | | | SAC | |
| Exp | osure | | | | <u> </u> |
| 10 | 10 Safety EX4 (XO) Listing of Exposure Data | | | | SAC |

| ICH | Listings | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title | | Title | Programming Notes | Deliverable<br>[Priority] |
| Adv | erse Events | | | | |
| 11 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 12 | Safety | CP_AE9<br>(XO) | Listing of All Adverse Events | | SAC |
| 13 | Safety | CP_AE9<br>(XO) | Listing of Drug Related Adverse Events | | SAC |
| 14 | Safety | CP_AE9a<br>(xo) | Listing of Serious Adverse Events | | SAC |
| 15 | Safety | CP_AE9 (xo) | Listing of Adverse Events Leading to<br>Permanent Discontinuation of Study<br>Treatment or Withdrawal from Study | | SAC |
| LAF | S | | ı , | | |
| 16 | Safety | CP_LB6 (xo) | Listing of Clinical Chemistry with Grade 2 or Higher Lab Abnormalities | Include all tests in which we have DAIDS criteria. | SAC |
| 17 | Safety | CP_LB6 (xo) | Listing of All Clinical Chemistry Laboratory Data for Subjects with Grade 2 or Higher Lab Abnormalities | Include all tests in which we have DAIDS criteria. | SAC |
| 18 | Safety | CP_LB6 (xo) | Listing of Hematology with Grade 2 or Higher Lab Abnormalities | Include all tests in which we have DAIDS criteria. | SAC |
| 19 | Safety | CP_LB6 (xo) | Listing of All Hematology Laboratory Data for Subjects with Grade 2 or Higher Lab Abnormalities | Include all tests in which we have DAIDS criteria. | SAC |
| 20 | Safety | UR2b | Listing of Urinalysis Data for Subjects with Positive Dipstick or Microscopic Results | | SAC |

| ICH | CH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | is | | | | |
| 21 | Safety | CP_EG4 (xo) | Listing of ECG Values of Potential Clinical Importance | | SAC |
| 22 | Safety | CP_EG4 (xo) | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance | | SAC |
| 23 | Safety | CP_EG6 (xo) | Listing of Abnormal ECG findings | | SAC |
| Vita | l Signs | | | | |
| 24 | Safety | CP_VS5<br>(XO) | Listing of Vital Signs of Potential Clinical Importance | | SAC |
| 25 | Safety | CP_VS5<br>(XO) | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

# 10.11.8. Non-ICH Listings

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / TST | | <b>Programming Notes</b> | Deliverable<br>[Priority] | |
| AE | | | | | |
| 26 | Safety | AE2 | Relationship between System Organ Class and<br>Verbatim Text | | SAC |
| PK | | | | | |
| 27 | PK Plasma<br>Concentration | pkcl1x | Listing of DTG Plasma Concentration-time Data | | SAC |
| 28 | 28 PK Plasma concentration pkcl1x | | Listing of 3TC Plasma Concentration-time Data | | SAC |
| 29 | PK Plasma Concentration pkpl1x | | Listing of DTC Plasma PK Parameters based on Actual Sampling Time | | SAC |
| 30 | PK Plasma<br>Concentration | pkpl1x | Listing of 3TC Plasma PK Parameters based on Actual Sampling Time | | SAC |
| 31 | PK Plasma<br>Concentration | pkpl1x | Listing of DTC Plasma PK Parameters based on Nominal Sampling Time | | SAC |
| 32 | PK Plasma<br>Concentration | pkpl1x | Listing of 3TC Plasma PK Parameters based on Nominal Sampling Time | | SAC |
| 33 | PK Parameter<br>BE Summary | mid20167,<br>listing 33 | Listing of Individual DTG Plasma PK Parameter Treatment Ratios based on Actual Sampling Time - Bioequivalence Assessment | | SAC |
| 34 | PK Parameter mid20167,<br>BE Summary listing 33 | | Listing of Individual 3TC Plasma PK Parameter Treatment Ratios based on Actual Sampling Time - Bioequivalence Assessment | | SAC |

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| 35 | PK Parameter<br>FD Summary | mid20167,<br>listing 33 | | SAC | |
| 36 | PK Parameter<br>FD Summary | mid20167,<br>listing 33 | Listing of Individual 3TC Plasma PK Parameter Treatment Ratios based on Actual Sampling Time – Food Effect | | SAC |
| 37 | 1 RH Summary Lighting 33 | | Listing of Individual DTG Plasma PK Parameter<br>Treatment Ratios based on Nominal Sampling Time -<br>Bioequivalence Assessment | | SAC |
| 38 | PK Parameter<br>BE Summary | mid20167,<br>listing 33 | Listing of Individual 3TC Plasma PK Parameter<br>Treatment Ratios based on Nominal Sampling Time -<br>Bioequivalence Assessment | | SAC |
| 39 | PK Parameter<br>FD Summary | mid20167,<br>listing 33 | Listing of Individual DTG Plasma PK Parameter Treatment Ratios based on Nominal Sampling Time – Food Effect | | SAC |
| 40 | PK Parameter mid /III6 / | | Listing of Individual 3TC Plasma PK Parameter Treatment Ratios based on Nominal Sampling Time – Food Effect | | SAC |
| 41 | PK Parameter BE Summary N/A RAW SAS Output from Statistical Analysis of Logetransformed DTG Plasma PK Parameters based on Actual Sampling Time - Bioequivalence Assessment | | | SAC | |
| 42 | PK Parameter<br>BE Summary N/A | | RAW SAS Output from Statistical Analysis of Loge-<br>transformed 3TC Plasma PK Parameters based on<br>Actual Sampling Time - Bioequivalence Assessment | | SAC |

| Non- | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 43 | PK Parameter<br>FD Summary | N/A I transformed DTG Plasma PK Parameters based on | | | SAC |
| 44 | PK Parameter FD Summary RAW SAS Output from Statistical Analysis of Logetransformed 3TC Plasma PK Parameters based on Actual Sampling Time - Food Effect | | | SAC | |
| 45 | PK Parameter N/A RAW SAS transformed | | RAW SAS Output from Statistical Analysis of Logetransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Bioequivalence Assessment | | SAC |
| 46 | PK Parameter RF Summary N/A RAW S transfor | | RAW SAS Output from Statistical Analysis of Loge-<br>transformed 3TC Plasma PK Parameters based on<br>Nominal Sampling Time - Bioequivalence Assessment | | SAC |
| 47 | 7 PK Parameter N/A RAW SAS Output f transformed DTG P | | RAW SAS Output from Statistical Analysis of Logetransformed DTG Plasma PK Parameters based on Nominal Sampling Time - Food Effect | | SAC |
| 48 | PK Parameter<br>FD Summary | N/A | RAW SAS Output from Statistical Analysis of Logetransformed 3TC Plasma PK Parameters based on Nominal Sampling Time - Food Effect | | SAC |

## 10.12. Appendix 12: Example Mock Shells for Data Displays

Example : PK\_T1

Protocol : 204994 Page 1 of n

Population : PK Parameter BE Summary (programming note: 'PK Parameter BE (or FD) Summary' depending each display in TOC)

### Table xx.xx

Summary of Statistical Analysis of Loge-transformed DTG Plasma Pharmacokinetic Parameters based on Actual Sampling Time

| Parameter | Comparison | Adjus | ted Geon | netric Mean | Ratio | 90% Confidence | %CVw |
|---|---|---|---|---|---|---|---|
| | Test vs Reference | n | Test | n Ref | (Test/Ref) | Interval for Ratio | |
| C <sub>max</sub> (units) | [Test treatment description] vs | | xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |
| $AUC_{(0-t)}(units)$ | [Reference treatment description] vs<br>[Test treatment description] vs<br>[Reference treatment description] | x | xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |
| $AUC_{(0-\infty)}(units)$ | | x | xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |
| C <sub>24</sub> (units) | [Test treatment description] vs<br>[Reference treatment description] | | xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |


Example : PK\_T2 Protocol : 204994

Population : PK Parameter BE Summary

### Table xx.xx

Summary of Statistical Analysis of Median Difference and Confidence Interval for DTG Pharmacokinetic Parameters based on Actual Sampling Time

| Parameter | Comparison | Median | D. C | Estimated Median Diff | 90% Confidence |
|---|---|---|---|---|---|
| | Test vs Reference | n Test<br> | n Ref<br> | (Test - Ref) | Interval for Diff |
| $T_{lag}(units)$ | [Test treatment description] vs<br>[Reference treatment description] | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) |
| $T_{max}$ )(units) | [Test treatment description] vs<br>[Reference treatment description] | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) |

Example :  $PK_F1$  Page 1 of n Protocol : 204994

Population : PK Parameter BE Summary

Figure xx.xx

Treatment Comparative Plot of Adjusted Geometric Mean (95% CI) with Individual Subjects

DTG Plasma Pharmacokinetic Parameters



Programming note: add footnote for treatment A, B.

204994

Example : PK\_F2 Page 1 of n

Protocol : 204994

Population : PK Parameter BE Summary

Figure xx.xx

Geometric Mean Treatment Ratio and 90% CI of DTG Plasma Pharmacokinetic Parameters



Note: The reference lines at ratios of 0.80, 1.25 represent BE criterion.

Programming note: add footnote for treatment A, B.

204994


Example: SAFE\_T1 Protocol: 204994

Population: Safety

Table xx.xx
Number of Subjects with Change from Baseline Vital Signs Category

| VSTEST | Pl. Time | Subject<br>Position | Flagging category | Test<br>(N=XX) | Reference (N=XX) |
|---|---|---|---|---|---|
| Diastolic Blood Pressure (mmHg) | Time 1 | Supine | n | XX | XX |
| . 5. | | | <pre>Increase &gt;=20</pre> | 0 | XX(XX%) |
| | | | <pre>Increase &gt;=40</pre> | XX(XX%) | 0 |
| | | | Decrease >=20 | 0 | XX(XX%) |
| | | | Decrease >=40 | XX (XX%) | 0 |
| | Time 2 | Supine | n | XX | XX |
| | | | Increase >=20 | 0 | XX (XX%) |
| | | | <pre>Increase &gt;=40</pre> | XX (XX%) | 0 |
| | | | Decrease >=20 | 0 | XX(XX%) |
| | | | Decrease >=40 | XX (XX%) | 0 |

204994


Example: SAFE\_L1 Protocol: 204994

Population: Screening

Listing X
Listing of Subjects Excluded from Analysis Populations

| Population | No. of<br>Subjects | No.<br>Subj<br>Excl | ects | Subject numbers |
|---|---|---|---|---|
| Screening | xxx | xx | ×××. | xxx, xxx, xxx. |
| Safety | xx | 0 | , | , |
| PK Plasma Concentration | XX | XX | XXX | |
| PK Parameter BE Summary | XX | XX | XXX | |
| PK Parameter Food Effect Summary | XX | XX | XXX | |


Example: PK\_T3
Protocol: 204994

Population: PK Plasma Concentration

Table x.xx
DTG Drug Concentration (unit) for the Test Formulation B

| ID Seq Period | 16.0<br>BLQ* |
|---|---|
| 0.0 0.33 0.66 1.0 1.5 2.0 3.0 4.0 6.0 8.0 12.0 | |
| A TR 14 May 0.00 BLQ* 52.01 95.03 122.20 77.88 65.15 46.24 19.20 14.99 BLQ* | BLQ* |
| B RT 21 May 0.00 BLQ* 56.66 80.85 102.00 86.41 63.81 49.20 24.00 11.37 8.24 | BLQ* |
| C RT 21 May 0.00 28.63 201.50 189.80 188.70 136.20 97.64 64.53 32.08 20.63 14.59 | BLQ* |
| E TR 14 May 0.00 BLQ* 9.04 34.32 47.70 52.79 59.47 32.61 17.61 8.76 BLQ* | BLQ* |
| F RT 21 May 0.00 BLQ+ 55.33 66.40 58.97 48.29 43.19 34.23 17.30 6.15 BLQ+ | BLQ* |
| G TR 14 May 0.00 BLQ* 33.15 45.64 54.19 34.13 32.78 21.73 10.75 8.35 BLQ* | BLQ* |
| H RT 21 May 0.00 35.38 79.14 100.90 70.71 48.43 30.73 26.19 8.65 6.83 BLQ* | BLQ* |
| I TR 14 May 0.00 BLQ* 64.57 76.52 89.51 86.21 69.04 50.96 21.55 13.71 7.55 | BLQ* |
| K RT 21 May 0.00 BLQ+ 79.34 99.41 154.80 58.60 57.12 32.57 19.82 BLQ+ BLQ+ | BLQ* |
| L TR 14 May 0.00 14.78 55.54 56.88 46.87 37.29 28.75 25.20 BLQ* BLQ* BLQ* | BLQ* |
| M TR 14 May 0.00 BLQ+ BLQ+ BLQ+ BLQ+ BLQ+ 8.37 23.15 19.74 16.49 5.74 | 5.18 |
| N RT 21 May 0.00 BLQ* 37.76 28.58 21.56 19.02 13.25 12.44 638 BLQ* BLQ* | BLQ* |
| O RT 21 May 0.00 BLQ+ 27.85 43.30 43.30 32.57 29.59 25.42 16.89 7.68 BLQ+ | BLQ* |
| P TR 14 May 0.00 BLQ+ 68.25 52.57 51.97 28.64 23.70 12.74 BLQ+ BLQ+ BLQ+ | BLQ* |
| Q RT 21 May 0.00 BLQ+ 5.90 13.00 27.54 13.32 12.34 9.81 9.73 BLQ+ BLQ+ | BLQ* |
| R TR 14 May 0.00 BLQ+ 18.92 35.77 53.93 60.43 47.44 41.72 16.66 8.87 5.49 | BLQ* |
| | : |
| MEAN 0.00 4.92 52.81 63.69 70.87 51.26 42.65 31.80 15.04 7.73 2.60 | 0.32 |
| STD 0.00 11.26 47.05 45.04 49.76 33.66 24.64 15.42 8.60 6.57 4.42 | 1.29 |
| CV 228.66 89.09 70.72 70.22 65.66 57.79 48.51 57.18 84.94 169.84 | 400 |

Lower limit of quantitation is 5 ng/mL. Any concentration below this limit is reported as Below Limit of Quantitation (BLQ) except at time 0. Zero is used in the calculation of area under the curve (AUC) for times preceding the first observed concentration and in the calculation of summary statistics.

204994


Example: PK\_T4
Protocol: 204994

Population: PK Plasma Concentration

| ID | Seq | Period | TEST FORMULATION | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Cmax<br>(ng/mL) | tmax<br>(h) | AUCT<br>(ng·h/mL) | AUCI<br>(ng·h/mL) | AUCT<br>(%) | ۱<br>(h <sup>n</sup> ) | TLIN<br>(h) | LQCT<br>(h) | t%<br>(h) |
| A | TR | 14 May | 122 | 1.50 | 365 | 409 | 89 | 0.3002 | 2.0 | 8.0 | 2.3 |
| В | RT | 21 May | 102 | 1.50 | 405 | 432 | 94 | 0.2384 | 3.0 | 12.0 | 2.9 |
| С | RT | 21 May | 202 | 0.66 | 703 | 774 | 91 | 0.1776 | 4.0 | 12.0 | 3.9 |
| Е | TR | 14 May | 59 | 3.00 | 233 | 256 | 91 | 0.3680 | 3.0 | 8.0 | 1.9 |
| F | RT | 21 May | 66 | 1.00 | 247 | 265 | 93 | 0.3902 | 3.0 | 8.0 | 1.8 |
| G | TR | 14 May | 54 | 1.50 | 178 | 205 | 87 | 0.2768 | 3.0 | 8.0 | 2.5 |
| Н | RT | 21 May | 101 | 1.00 | 246 | 263 | 94 | 0.3437 | 2.0 | 8.0 | 2.0 |
| I | TR | 14 May | 90 | 1.50 | 408 | 433 | 94 | 0.2486 | 3.0 | 12.0 | 2.8 |
| K | RT | 21 May | 155 | 1.50 | 315 | 372 | 85 | 0.3379 | 3.0 | 6.0 | 2.1 |
| L | TR | 14 May | 57 | 1.00 | 140 | 331 | 42 | 0.1318 | 3.0 | 4.0 | 5.3 |
| М | TR | 14 May | 23 | 4.00 | 165 | 195 | 85 | 0.1485 | 6.0 | 16.0 | 4.7 |
| N | RT | 21 May | 38 | 0.66 | 88 | 113 | 78 | 0.2620 | 2.0 | 6.0 | 2.6 |
| 0 | RT | 21 May | 43 | 1.00 | 183 | 215 | 85 | 0.2671 | 3.0 | 8.0 | 2.6 |
| р | TR | 14 May | 68 | 0.66 | 122 | 148 | 83 | 0.5031 | 1.5 | 4.0 | 1.4 |
| Q | RT | 21 May | 28 | 1.50 | 68 | 113 | 60 | 0.1833 | 1.5 | 6.0 | 3.8 |
| R | TR | 14 May | 60 | 2.00 | 275 | 292 | 94 | 0.2546 | 3.0 | 12.0 | 2.7 |
| | 1 | | S | | 51<br>13<br>13<br>14 | | | | | | |
| MEAN* | 20 | 586 | 79 | 1.50 | 259 | 301 | 84 | 0.2770 | 3.0 | 8.0 | 2.8 |
| STD | | C 1050 | 48 | 0.89 | 158 | 164 | 14 | 0.0967 | 1.1 | 3.3 | 1.1 |
| cv | 201 | 88488 | 61 | 59.35 | 61 | 54 | 17 | 34.92 | 37.3 | 38.5 | 37.9 |

Example: PK\_T5
Protocol: 204994

Protocol: 204994 Page 1 of n

Population: PK Parameter BE Summary

Table x.xx

DTG Parameter Analysis - Data based on Actual Time - Bioequivalence Assessment

| | | Raw Scale | Log Scale | | |
|---|---|---|---|---|---|
| Ð | Test<br>AUCT | Reference<br>AUCT | Relative<br>AUCT (%) | Test<br>ln(AUCT) | Reference<br>ln(AUCT) |
| A | 365 | 375 | 97 | 5.8998 | 5.9269 |
| В | 405 | 595 | 68 | 6.0038 | 6.3885 |
| С | 703 | 471 | 149 | 6.5553 | 6.1548 |
| E | 233 | 190 | 123 | 5.4510 | 5.2470 |
| F | 247 | 257 | 96 | 5.5093 | 5.5490 |
| G | 178 | 175 | 102 | 5.1817 | 5.1647 |
| н | 246 | 382 | 65 | 5.5053 | 5.9454 |
| I | 408 | 361 | 113 | 6.0112 | 5.8888 |
| K | 315 | 218 | 144 | 5.7525 | 5.3844 |
| L | 140 | 92 | 153 | 4.9416 | 4.5217 |
| М | 165 | 269 | 61 | 5.1059 | 5.5947 |
| N | 88 | 106 | 83 | 4.4773 | 4.6634 |
| 0 | 183 | 290 | 63 | 5.2094 | 5.6698 |
| P | 122 | 230 | 53 | 4.8040 | 5.4380 |
| Q | 68 | 144 | 47 | 4.2195 | 4.969\$ |
| R | 275 | 344 | 80 | 5.6167 | 5.8406 |
| : | | | : | : | |
| MEAN | 259 | 281 | 94 | 5.3903 | 5.5217 |
| STD | 158 | 136 | 35 | 0.61 | 0.52 |
| cv | 61 | 48 | 37 | | - |